CLINICAL TRIAL: NCT06003322
Title: Non - Incised Papilla Versus Single Flap Technique In The Reconstruction Of Intrabony Defect: a Randomized Controlled Trial
Brief Title: Non - Incised Papilla Versus Single Flap Technique In The Reconstruction Of Intrabony Defect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Assiut University (Other); Egyptian Russian University (Network)
Responsible Party: Principal Investigator, Alaa Talaat Ali, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER243
Record Dates: First submitted 2023-06-24; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Periodontal Attachment Loss
MeSH Terms: conditions — Periodontal Attachment Loss

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non - Incised Papilla surgical approach NIPSA for intrabony defect (Experimental): Group I will be allocated to non - Incised Papilla surgical approach NIPSA for intrabony defect with DBBM and PRF
  Interventions: Procedure: non - Incised Papilla surgical approach NIPSA for intrabony defect
- single-flap approach (Active Comparator): group II will be allocated to single-flap approach SFA for intrabony defect with DBBM and PRF
  Interventions: Procedure: single-flap approach SFA

INTERVENTIONS:
Procedure: non - Incised Papilla surgical approach NIPSA for intrabony defect — As described by Rodríguez and Caffesse in 2018, a single incision apical to the defect ,on the buccal aspect, only one apical horizontal or oblique incision will be made in the alveolar mucosa, as far removed as possible from the interdental papillae and marginal keratinized tis- sues.
  Following flap reflection, the bony defect will be examined carefully. Root planing is performed,. Flap closure will be performed by horizontal mattress sutures, placed 3 mm away from the borders, will be used as the first line of closure, promoting connective tissue contact between both edges of the incision, and single interrupted sutures will then be placed as a second line of closure. Using 5/0 polypropylene monofilament suture, Assut, Swiss
  Arms: non - Incised Papilla surgical approach NIPSA for intrabony defect
Procedure: single-flap approach SFA — As described by Trombelli et al 2010, A horizontal, butt-joint incision will be performed at the interdental papilla 1-2 mm coronal to the bone crest (as detected through pre-operative bone sounding).
  -A buccal mucoperiosteal envelope flap will be elevated by using a microsurgical periosteal elevator, leaving the residual portion of the interdental supracrestal soft tissues undetached.Flap closure will be performed by a horizontal internal mattress suture,will be performed at the base of the papilla, and a second internal mattress suture (vertical or horizontal) was performed between the most coronal portion of the flap and the most coronal portion of the palatal/lingual papilla. Using a resorbable suture
  Arms: single-flap approach

SUMMARY:
The present study will aim to assess the effectiveness of the non-Incised Papilla surgical approach NIPSA used for the surgical debridement of deep intraosseous defects compared to the single-flap approach SFA.

Primary outcome: interproximal clinical attachment level gain Secondary outcomes: residual probing pocket depth (PPD), pocket depth (PD) reduction, recession (REC), location of the tip of the papilla (TP), width of the keratinized tissue (KT), wound closure (WC), supra-alveolar attachment gain (SUPRA-AG)

DETAILED DESCRIPTION:
The present study will aim to assess the effectiveness of the non-Incised Papilla surgical approach NIPSA used for the surgical debridement of deep intraosseous defects compared to the single-flap approach SFA.

Primary outcome: interproximal clinical attachment level gain Secondary outcomes: residual probing pocket depth (PPD), pocket depth (PD) reduction, recession (REC), location of the tip of the papilla (TP), width of the keratinized tissue (KT), wound closure (WC), supra-alveolar attachment gain (SUPRA-AG)

ELIGIBILITY:
Inclusion Criteria:

* - Age > 18 years
* Diagnosis with stage III-IV periodontitis.
* Presence of one or more intrabony defects with probing pocket depth (PPD) > 5 mm and radiographic defect depth > 4 mm.
* Full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) < 30% (measured at four sites per tooth).
* No relevant systemic condition or disease.

Exclusion Criteria:

Third molars and teeth with type III mobility or with an incorrect endodontic or restorative treatment.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-08-07 (Estimated); Study Completion 2024-09-07 (Estimated)

PRIMARY OUTCOMES:
interproximal clinical attachment level change | at baseline ,6 and 12 months
  CAL, measured in the interproximal space from the CEJ to the base of the pocket(BP)using a millimeter periodontal probe

SECONDARY OUTCOMES:
residual probing pocket depth (PPD), pocket depth (PD) change, | at at baseline ,6 and 12 months
  -Inter- proximal PD, measured in the interproximal space from the gingival margin to the BP measured by a millimeter periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: ALAA T ALI, PhD, Study Director — Assiut University
Locations (1):
- faculty of dentistry ,Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No